CLINICAL TRIAL: NCT06156319
Title: A Multicentre Cohort Study on the Effect of Clonal Hematopoiesis on Prognosis in Patients With Myocardial Infarction Based on Residual Inflammation Risk
Brief Title: Clonal Hematopoiesis on Prognosis in Patients With Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yang Jing (Other)
Responsible Party: Sponsor-Investigator, Yang Jing, physician, Chongqing Emergency Medical Center
Organization: Chongqing Emergency Medical Center (Other)
Other Study IDs: 2023MSXM019
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: To Investigate the Effect of CHIP on Renal Insufficiency in AMI Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: CHIP group: Patients diagnosed with AMI combined with CKD stage II-IV underwent PCI and were identified as CHIP carriers by gene targeted sequencing.
  Non-chip group: Patients diagnosed with AMI combined with CKD stage II-IV underwent PCI and were identified as non-CHIP carriers by gene targeted sequencing.
  Interventions: Other: No intervention
- Group 2: CHIP group: Patients diagnosed with AMI combined with ESRD underwent PCI and were identified as CHIP carriers by gene targeted sequencing Non-chip group: Patients diagnosed with AMI combined with ESRD underwent PCI and were identified as non-CHIP carriers by gene targeted sequencing
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is an observational study without intervention. It is planned to include 500 patients with AMI from October 2023 to July 2026.The study was divided into three parts. Part I: To investigate the effect of CHIP on renal insufficiency in AMI patients.

Part two: To investigate the effect of CHIP on cardiovascular outcomes in patients with AMI complicated with CKD stage II-IV nephropathy. Part three: To investigate the effects of CHIP on cardiovascular and renal outcomes in AMI patients with ESRD. Study endpoint: Primary end points: all-cause death, cardiac death, and nonfatal myocardial infarction. Secondary endpoints: angina pectoris requiring hospitalization, nonfatal stroke, and nonfatal heart failure.

DETAILED DESCRIPTION:
This is an observational study without intervention. It is planned to include 500 patients with AMI from October 2023 to July 2026.The study was divided into three parts. Part I: To investigate the effect of CHIP on renal insufficiency in AMI patients.

Patients with confirmed AMI were divided into two groups based on eGFR values:

AMI+ normal renal function group (eGFR≥90 ml/min); AMI+ renal dysfunction group (eGFR < 90 ml/min). Main outcome measures: CHIP carrying frequency, expression levels of IL-1β, IL-6, CRP, TNF-α, NLRP3 and other inflammatory factors.

Part two: To investigate the effect of CHIP on cardiovascular outcomes in patients with AMI complicated with CKD stage II-IV nephropathy. Patients with confirmed AMI complicated with CKD stage II-IV were divided into two groups according to CHIP sequencing results: CHIP group: Patients diagnosed with AMI combined with CKD stage II-IV underwent PCI and were identifi ed as CHIP carriers by gene targeted sequencing. Non-chip group: Patients diagnosed with AMI combined with CKD stage II-IV underwent PCI and were identified as non-CHIP carriers by gene targeted sequencing. Study endpoint: Primary endpoints: all-cause death, cardiac death, nonfatal myocardial infarction,50% decrease in eGFR, or ESKD. Secondary endpoints: angina pectoris requiring hospitalization, nonfatal stroke, and nonfatal heart failure. Part III: To investigate the effects of CHIP on cardiovascular and renal outcomes in AMI patients with ESRD. Patients with confirmed AMI combined with ESRD were divided into two groups according to CHIP sequencing results: CHIP group: Patients diagnosed with AMI combined with ESRD underwent PCI and were identified as CHIP carriers by gene targeted sequencing. Non-chip group: Patients diagnosed with AMI combined with ESRD underwent PCI and were identified as non-CHIP carriers by gene targeted sequencing. Study endpoint: Primary end points: all-cause death, cardiac death, and nonfatal myocardial infarction. Secondary endpoints: angina pectoris requiring hospitalization, nonfatal stroke, and nonfatal heart failure.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with AMI received PCI.

Exclusion Criteria:

patients with severe heart disease, severe liver and kidney insufficiency, pregnancy, etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosing patients with AMI.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
MACE | 2 years
  all-cause death, cardiac death, and nonfatal myocardial infarction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang Z, Li Y, Yan C, Zhang X, Zhang Q, Li J, Tian X, Qiu M, Liang Z, Ma S, Na K, Li Z, Chen S, Zhao Y, Qi Z, Liu X, Han Y. Clonal hematopoiesis of indeterminate potential in patients with acute coronary syndrome undergoing percutaneous coronary intervention in the absence of traditional risk factors. Clin Res Cardiol. 2023 Apr;112(4):506-517. doi: 10.1007/s00392-022-02039-6. Epub 2022 Jun 15. PMID 35704087